CLINICAL TRIAL: NCT03074890
Title: Observational Study to Assess the Safety and Clinical Effectiveness of the Hospital Universitario de Canarias Massive Transfusion Protocol
Brief Title: Evaluating of the Hospital Universitario de Canarias Massive Transfusion Protocol
Acronym: PHM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Principal Investigator, María del Carmen Martín Lorenzo, Dr, Hospital Universitario de Canarias
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TRAMA-05-2014
Record Dates: First submitted 2016-12-22; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Massive Transfusion; Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (cases) (Experimental): Intervention: Massive transfusion protocol resuscitation aiming at ratio 1:1:1 of blood components (RBC:FFP:PLT) and conventional coagulation tests guiding further resuscitation with blood products and procoagulant factors
  Interventions: Device: Application Protocol
- No Intervention (control)) (No Intervention): all patients with massive haemorrhage in which the massive transfusion protocol didn´t apply

INTERVENTIONS:
Device: Application Protocol — Application lMassive Transfusion Protocol
  Arms: Intervention (cases)

SUMMARY:
Massive haemorrhage is defined as the necessity of 3 or more packed red blood cells in one hour, the transfusion of 10 packed blood cells, the loss of the half of the blood volume, the loss of 4-5 cc/kg/h or more, and haemorrhage shock.

Haemorrhage shock provokes changes in the bloodstream with celular and organic disfunction. In many cases massive transfusion is needed to stabilize the vital function. This massive transfusion can have serious side effects (infectious and immunologic and no immunologic reactions) and increase the morbidity and mortality.

Massive transfusion protocols improve the survival in severe trauma injury patients. The transfusion of fixed rate of packed red blood cells, fresh frozen plasma and platelet concentrates have decreased the severity of trauma induced coagulopathy.

Recently several studies have shown the benefit of massive transfusion protocols with high transfusion ratios (1:1:1 RBC:FFP:PLT) in mortality after severe trauma. So early and aggressive transfusion improve the outcomes and the resources.

Massive Transfusion Protocol have been elaborated in the Hospital Universitario de Canarias with high transfusion ratios (1:1:1 RBC:FFP:PLT) . The goals of this protocol is to reduce the variability in the clinic experience, to reduce the transfusion necessities and to assure an safe treatment with blood products.

So with this study the investigators will evaluate if the goals of this Protocol are followed and if the use of this Protocol is really safe and efficient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with massive haemorrhage and surgery
* Informed consent

Exclusion Criteria:

* <18 years old patients
* Patients didn´t want to participate in this study
* Patients were participated in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
30-day Mortality | First 30 day after massive transfusion
Time to Hemostasis | admission to hospital discharge or 30 days, whichever comes first
  Time to hemostasis refers to the time that the subject achieved hemorrhage control (anatomic hemostasis and resuscitation complete)following emergency department arrival.

SECONDARY OUTCOMES:
Incidence of Massive Transfusion Related Serious Adverse Events | 30 days
  Immunological reactions No immunological reactions
Severity of coagulopathy associated with high transfusion ratios | 30 days post admission
Amount of Blood Products Given to Hemostasis | 24 hours from randomization
Amount of Blood Products Given From Hemostasis to 24 Hours After | 24 hours after admission

CONTACTS AND LOCATIONS:
Overall Officials: Vanesa González Fariña, MD, Principal Investigator — Hospital Universitario de Canarias; Juan J Jiménez Rivera, MD, Study Director — Hospital Universitario de Canarias; José M Raya Sánchez, MD, Study Director — Hospital Universitario de Canarias
Locations (1):
- Complejo Universitario de Canarias, Laguna del Marquesado, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spahn DR, Cerny V, Coats TJ, Duranteau J, Fernandez-Mondejar E, Gordini G, Stahel PF, Hunt BJ, Komadina R, Neugebauer E, Ozier Y, Riddez L, Schultz A, Vincent JL, Rossaint R; Task Force for Advanced Bleeding Care in Trauma. Management of bleeding following major trauma: a European guideline. Crit Care. 2007;11(1):R17. doi: 10.1186/cc5686. PMID 17298665
- [Background] Malone DL, Hess JR, Fingerhut A. Massive transfusion practices around the globe and a suggestion for a common massive transfusion protocol. J Trauma. 2006 Jun;60(6 Suppl):S91-6. doi: 10.1097/01.ta.0000199549.80731.e6. PMID 16763487
- [Background] Borgman MA, Spinella PC, Perkins JG, Grathwohl KW, Repine T, Beekley AC, Sebesta J, Jenkins D, Wade CE, Holcomb JB. The ratio of blood products transfused affects mortality in patients receiving massive transfusions at a combat support hospital. J Trauma. 2007 Oct;63(4):805-13. doi: 10.1097/TA.0b013e3181271ba3. PMID 18090009
- [Background] Leal-Noval SR, Munoz M, Asuero M, Contreras E, Garcia-Erce JA, Llau JV, Moral V, Paramo JA, Quintana M; Spanish Society of Anaesthesiology and Reanimation (SEDAR); Spanish Society of Haematology and Haemotherapy (SEHH); Spanish Society of Hospital Pharmacy (SEFH); Spanish Society of Intensive Care, Critical and Coronary Units (SEMICYUC); Spanish Society of Thrombosis and Haemostasis (SETH); Spanish Society of Blood Transfusion (SETS). [2013: The Seville document on consensus on the alternatives to allogenic blood transfusion. Update to the Seville document. Spanish Societies of Anaesthesiology (SEDAR), Haematology and Haemotherapy (SEHH), Hospital Pharmacy (SEFH), Critical Care Medicine (SEMICYUC), Thrombosis and Haemostasis (SETH) and Blood Transfusion (SETS)]. Farm Hosp. 2013 May-Jun;37(3):209-35. doi: 10.7399/FH.2013.37.3.133. Spanish. PMID 23789799
- [Background] Cotton BA, Au BK, Nunez TC, Gunter OL, Robertson AM, Young PP. Predefined massive transfusion protocols are associated with a reduction in organ failure and postinjury complications. J Trauma. 2009 Jan;66(1):41-8; discussion 48-9. doi: 10.1097/TA.0b013e31819313bb. PMID 19131804